CLINICAL TRIAL: NCT01882504
Title: An Open-label, Proof of Concept Study of Gevokizumab in the Treatment of the Acute, Inflammatory Phase of Pyoderma Gangrenosum
Brief Title: Proof of Concept Study of Gevokizumab in the Treatment of Pyoderma Gangrenosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X052170
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Pyoderma Gangrenosum
Keywords: Pyoderma Gangrenosum; Classic Pyoderma Gangrenosum; Atypical Pyoderma Gangrenosum; Peristomal Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — gevokizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gevokizumab (Experimental): Solution for subcutaneous injection
  Interventions: Drug: gevokizumab

INTERVENTIONS:
Drug: gevokizumab

SUMMARY:
The study will evaluate the safety and biologic activity of gevokizumab in subjects in the acute inflammatory phase of pyoderma gangrenosum.

ELIGIBILITY:
Inclusion Criteria:

* An established diagnosis of pyoderma gangrenosum
* Currently experiencing an inflammatory episode of pyoderma gangrenosum
* Contraceptive measures adequate to prevent pregnancy during the study

Exclusion Criteria:

* Clinical evidence of acutely infected pyoderma gangrenosum
* History of allergic or anaphylactic reactions to monoclonal antibodies
* History of recurrent or chronic systemic infections
* Female subjects who are pregnant, planning to become pregnant, have recently delivered, or are breast-feeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Improvement in the Investigator's Assessment of the pyoderma gangrenosum target ulcer | Day 1 through Day 84

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Miami, Florida
  - Miami Shores, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Verona, New Jersey
  - New York, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Knoxville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia